CLINICAL TRIAL: NCT03779360
Title: Investigating Anti-inflammatory Effects of Topical Antibiotics in an LPS Skin Challenge Model
Brief Title: Intradermal LPS and Antibiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Human Drug Research, Netherlands (Other)
Collaborators: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: CHDR1752-B
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Inflammation; Skin
MeSH Terms: conditions — Dermatitis | interventions — Erythromycin; Clindamycin; Prednisolone; Clobetasol; Dosage Forms; Lipopolysaccharides

STUDY DESIGN:
Intervention Model Description: An interventional, open-label, comparator controlled study to investigate the immunomodulatory effects of erythromycin and clindamycin in an LPS skin challenge model in healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjects 1-6 (Active Comparator): 7 day treatment of erythromycin and clindamycin twice daily on indicated skin areas prior to Clobetasol treatment; randomized either on the left or right arm for 2 days.
  Interventions: Drug: Erythromycin 4% topical gel formulation:; Drug: Clindamycin 1% lotion formulation:; Drug: Clobetasol propionate 0.05% topical formulation (crossover comparison):
- Subjects 7-24 (Experimental): 7 day treatment of erythromycin and clindamycin twice daily on indicated skin area prior to 4 Lipopolysaccharide injections and Clobetasol treatment; randomized either on the left or right arm for 2 days.
  Interventions: Drug: Erythromycin 4% topical gel formulation:; Drug: Clobetasol propionate 0.05% topical formulation (crossover comparison):; Other: Lipopolysaccharide
- Subjects 25-30 (Active Comparator): 0.5mg/kg prednisolone two days prior to Lipopolysaccharide injections
  Interventions: Drug: Prednisolone tablet (0.5mg/kg; parallel comparison):; Other: Lipopolysaccharide

INTERVENTIONS:
Drug: Erythromycin 4% topical gel formulation: — 7 day pre-treatment with erythromycin and clindamycin applied twice daily on marked area on left (erythromycin) and right side (clindamycin) of the volar lower arm. Erythromycin is a bacteriostatic antibiotic that belongs to the macrolide group of antibiotics. Macrolides act as bacteriostatic by reversibly binding to the P site on the 50S subunit of bacterial ribosomes. A topical gel formulation with hyprolose and ethanol.
  Arms: Subjects 1-6; Subjects 7-24
Drug: Clindamycin 1% lotion formulation: — 7 day pre-treatment with erythromycin and clindamycin applied twice daily on marked area on left (erythromycin) and right side (clindamycin) of the volar lower arm. Clindamcin is a bacteriostatic antibiotic that belongs to the lincosamide group of antibiotics. Lincosamides act as bacteriostatic by reversibly binding to the P site on the 50S subunit of bacterial ribosomes. A topical lotion formulation with ethanol.
  Arms: Subjects 1-6
Drug: Prednisolone tablet (0.5mg/kg; parallel comparison): — 2 day pre-treatment with prednisolone daily dose 0.5mg/kg (0.25mg/kg in the morning and 0.25mg/kg in the evening). Prednisolone tablet (0.5mg/kg; parallel comparison): Prednisolone is a synthetic corticosteroid with predominant glucocorticoid activity and as such it is widely used in the treatment for inflammatory and autoimmune diseases. Prednisolone exerts its effect by binding to cytoplasmic glucocorticoid receptors and subsequently activates glucocorticoid receptor mediated gene expression. This results in synthesis of certain anti-inflammatory proteins, while inhibiting the synthesis of certain inflammatory mediators.
  Arms: Subjects 25-30
Drug: Clobetasol propionate 0.05% topical formulation (crossover comparison): — 2 day pre-treatment with clobetasol propionate 0.05% topical formulation applied twice daily on marked area on left or right side of the volar lower arm.
  Clobetasol propionate 0.05% topical formulation (crossover comparison):
  Clobetasol propionate is a potent synthetic corticosteroid with anti-inflammatory, anti-pruritic, and vasoconstrictive properties. Clobetasol propionate exerts its effect by binding to cytoplasmic glucocorticoid receptors and subsequently activates glucocorticoid receptor mediated gene expression. This results in synthesis of certain anti-inflammatory proteins, while inhibiting the synthesis of certain inflammatory mediators. Specifically, clobetasol propionate appears to induce phospholipase A2 inhibitory proteins, thereby controlling the release of the inflammatory precursor arachidonic acid from membrane phospholipids by phospholipase A2.
  Arms: Subjects 1-6; Subjects 7-24
Other: Lipopolysaccharide — As TLR4 agonist, purified lipopolysaccharide prepared from Escherichia Coli: 113: H10:K negative (U.S. Standard Reference Endotoxin) will be used. This LPS batch is manufactured in the US by the National Institute of Health (NIH). Subjects will receive two intradermal doses of LPS in each forearm on day 0 (4 LPS injections in total, except for subjects 1-6 who receive none and subjects 25-27 will receive 2 LPS injections, only in the right arm). The dose per injection is 10 ng.
  Other Names: LPS
  Arms: Subjects 25-30; Subjects 7-24

SUMMARY:
Erythromycin and clindamycin are believed to have anti-inflammatory aspects. This study investigates the possible anti-inflammatory effects of erythromycin and clindamycin.

DETAILED DESCRIPTION:
Convincing mechanistic reports on the immunomodulatory action of erythromycin and clindamycin are scarce, rarely based on experiments in freshly isolated human immune cells, and potentially contradicting. Moreover, direct immunomodulatory effects of both antibiotics have never been demonstrated in vivo. The Centre for Human Drug Research Biomarker lab has studied in depth the immunomodulatory actions of erythromycin and clindamycin in vitro. These in vitro experiments on primary human immune cells demonstrated that both erythromycin and clindamycin are able to modulate the immune response of peripheral blood mononuclear cells upon stimulation with different immune triggers such as lipopolysaccharide (LPS) and polyI:C. In this current study the in vitro work will be translated to an in vivo study where it will be made into an intradermal LPS skin challenge model in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects, 18 to 45 years of age, inclusive. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, blood serology and urinalysis;
2. Body mass index (BMI) between 18 and 30 kg/m2, inclusive, and with a minimum weight of 50 kg;
3. Fitzpatrick skin type I-III (Caucasian);
4. Able and willing to give written informed consent and to comply with the study restrictions.
5. Able to work with the eDiary app.

Exclusion Criteria:

1. Any disease associated with immune system impairment, including auto-immune diseases, HIV and transplantation patients;
2. Type 1 or type 2 diabetes mellitus;
3. Any vaccination within the last 3 months;
4. Family history of psoriasis;
5. History of pathological scar formation (keloid, hypertrophic scar);
6. Have any current and / or recurrent pathologically, clinical significant skin condition at the treatment area (i.e. atopic dermatitis);
7. Hypersensitivity for dermatological marker at screening;
8. Requirement of immunosuppressive or immunomodulatory medication within 30 days prior to enrollment or planned to use during the course of the study;
9. Excessive sun exposure or a tanning booth within 3 weeks of enrollment;
10. Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times a year;
11. Loss or donation of blood over 500 mL within three months prior to screening. Or the donation of plasma within 14 days prior to screening;
12. Current smoker and/or regular user of other nicotine-containing products (e.g., patches);
13. History of or current drug or substance abuse considered significant by the PI (or medically qualified designee), including a positive urine drug screen.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-02-23 (Actual); Study Completion 2019-02-23 (Actual)

PRIMARY OUTCOMES:
Change in perfusion by Laser speckle contrast imaging (LSCI) | Baseline, 3, 6, 10, 24 and 48 hours post LPS injection
  Cutaneous microcirculation between pre and post-dose will be assessed using the laser speckle imager.
Change in erythema by Antera 3D camera and 2D camera | Baseline, 3, 6, 10, 24 and 48 hours post LPS injection
  Standardized photographs will be taken using the Antera camera (Antera 3D, Miravex, Ireland).
Change in erythema by clinical evaluation (erythema grading scale) | Baseline, 3, 6, 10, 24 and 48 hours post LPS injection
  At the specific time points pre and post dose the colour of the injected area is scored (erythema index), on a 4 point scale; normal, mild, moderate, severe.
Change in temperature by thermography in celsius | Baseline, 3, 6, 10, 24 and 48 hours post LPS injection
  Skin temperature will be measured using a thermal imaging camera.
Change in skin microbiome | Baseline, 3, 6, 10, 24 and 48 hours post LPS injection
  Collection of skin culture samples is a non-invasive procedure where a sterile polyester flock tip per site is passed along the surface of treated and non-treated areas.
  bacteria studied include but are not limited to: Acinetobacter Anaerococcus Corynebacterium Enhydrobacter Finegoldia Lactobacillus Micrococcus Paracoccus Peptoniphilus Prevotella Propionibacterium Staphylococcus Streptococcus

CONTACTS AND LOCATIONS:
Overall Officials: Matthijs Moerland, PhD, Principal Investigator — Researc Director
Locations (1):
- Centre for Human Drug Research, Leiden, South Holland, Netherlands